CLINICAL TRIAL: NCT00425295
Title: Effectiveness of Human Simulation Training for Medical Crisis Management Skills
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: too much cross over bias between small numbers of participants
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Lillian Emlet, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 0501050
Record Dates: First submitted 2007-01-19; First posted 2007-01-22 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Behavioral: Human Simulation Training
- 2 (Experimental)
  Interventions: Behavioral: Human Simulation Training

INTERVENTIONS:
Behavioral: Human Simulation Training — Fellows will undergo Human Simulation Training (HST) composed of one 1 hour session of high-fidelity simulation of crisis scenarios requiring management of critical care skills, including triage, Advanced Cardiac Life Support (ACLS), team management, and difficult airway management.

SUMMARY:
The main purpose of this study is to assess the effectiveness of human simulation in the training of the leadership, cognitive, and psychomotor skills required to lead medical crisis management teams. All participants in the study are trainees in the University of Pittsburgh Medical Center (UPMC) Multi-Disciplinary Critical Care Training Program (MCCTP.) All trainees will have received the standard critical care medicine-training curriculum including basic airway management, management of hypotension, unstable cardiac arrhythmias, difficult airway management and crisis team training. The participants will have also completed six months of baseline clinical training, which includes responding to medical emergencies at UPMC.

The specific aims of this study are:

1. To assess the effectiveness of Human Simulation Training (HST) as an educational tool for teaching medical crisis management.
2. To determine the effect of HST on objective measures of performance in the domains of communication, leadership, cognition and psychomotor skills.

DETAILED DESCRIPTION:
The use of Medical Emergency Teams (METS) for handling in-hospital medical crisis decreases mortality and improves patient safety. Adverse in-hospital events occur in about 4-17% of hospital admissions. Of these, 70% are thought to be preventable. The most serious adverse in-hospital event is unexpected cardiac arrest which carries a mortality rate of 50-80% [1]. One approach to reducing this adverse event is the use of METS. Unlike traditional cardiopulmonary resuscitation teams, which respond to cardiac arrests, METS respond to medical crises early on and aim to prevent the progression of problems into unstable situations. The implementation of METS have been found to decrease the number of unexpected cardiac arrests, intensive care unit transfers and in-hospital mortality [1]. Bellomo et al. further found that the implementation of a MET not only decreases hospital mortality but also decreases incidence of post-operative complications [2]. As an integral part of the MET, a critical care physician must have the communication and leadership skills to effectively manage the team, the cognitive skills to adequately assess/judge the situation and guide plan of actions, and the psychomotor skills to perform necessary procedures.

Existing methods for teaching medical crisis management are inadequate. The instruction of medical trainees in the management of acute medical crisis is often done through didactic teaching, problem based learning, and apprenticeship. It is not uncommon for a trainee's first experience managing medical crisis to be on a real patient who is experiencing a real medical crisis with significant consequences. This form of training is limited and clearly sub-optimal for many reasons. Didactic training and problem based learning may be useful in instilling medical knowledge but is often inadequate in teaching the communication skills and critical thinking that is involved in managing medical crises. Further, the urgency and complexity of medical crisis is not well understood without first-hand experience. In general, although medical crises are relatively common, trainees get limited opportunities for the repetition required to hone their management skills. Some medical crises, such as respiratory distress with difficult airway, are extremely rare and will not often be experienced by most trainees. Moreover, when they do occur, trainees may not have enough supervision and hence do not receive appropriate feedback. Thirdly, clinical apprenticeship does not provide for standardization of training and feedback for the trainees. Lastly, most trainees are not allowed to view the consequences of the errors made while managing medical crises as most supervisors will intervene to prevent patient injury or harm [3-6].

HST can be used as an educational tool for teaching medical crisis management. Simulation training has been used in other fields, such as aviation and the military, to train people to do complex tasks with potentially dangerous consequences [7-13]. A curriculum using HST may be a useful at surpassing some of the limitations of traditional training noted above[14]. The full body human simulator such as Laerdal's Sim Man, can be programmed to present a wide range of physiologic conditions and physical exam findings. Using this human simulator, a wide variety of medical crises can be programmed to recreate real-life situations. The human simulator also allows the re-creation of clinically important but rare situations. The human simulator will also allow trainees to manage medical crises repetitively until a satisfactory level of proficiency can be reached.

Most importantly, HST allows trainees to repetitively experience dangerous situations and practice their crisis management skills. Trainees can now benefit by seeing their management errors run their course without placing patients at risk. HST allows for providing immediate feedback. This technology is portable and hence allows for trainees from various institutions within a particular region to have standardized training and feedback. The 1999 Institute of Medicine Report, "To Err is Human," challenged the medical community to confront the issue of medical error. One innovative approach that was mentioned for performance improvement and healthcare training was the use of human simulators [15].

Human Simulators are a valuable and valid performance evaluation tool. Human simulators have long been used in the field of medicine for evaluation. In particular, the field of anesthesia has taken the lead in terms of using advanced full body simulators for resident and physician training and evaluation. Instructors in the field of anesthesia have used human simulators to re-create dangerous and complex intra-operative crises to help their trainees acquire, test, and practice skills of crisis resource management without placing patients at risk [16-18]. By using evaluation techniques such as videotaped review and checklists, anesthesia instructors have been able to assess the behavioral and technical performances of trainees[18-21].

The effectiveness of HST as a training tool in medical crisis management needs to be explored.

Due to the success of human simulation as an educational tool for anesthesia crisis, HST is now being used as a tool for training medical emergency teams for dealing with medical crisis. Lighthall et al. has showed that HST can be used to teach crisis management to internal medicine residents[22]. This study showed that the majority of participants felt that simulator training had an educational value, but did not quantify their performance of technical and non-technical skills. DeVita et al. looked at the effect of HST on improving crisis team skills. This study found that repeated experience using the simulator with immediate feedback improved team performance in terms of correctly completing the steps necessary for patient/simulator survival[23]. There are no studies, which look at whether HST improves crisis management skills in a randomized study design.

2.2 Significance The field of simulation education is highly evolved in other high-risk industries such as aviation and nuclear power plants. Its time is coming in medical education, particularly with the emerging emphasis on improved patient safety. Proven and practical outcome based educational programs are needed to support the cultural changes necessary to influence the changes in fields of education in clinically relevant domains such as medical crisis resource management.

Medical crisis management skills are essential to the function of METS. HST is a useful tool that can safely re-create medical crises to teach and evaluate trainees in these skills. Although HST has been widely studied in anesthesia crisis management, there are no studies that look at the effect of HST on medical crisis management skills. We feel that this study will help to determine what effect if any, HST has on the communication, leadership, cognitive and psychomotor skill level needed to be effective at medical crisis management.

The participants for this prospective, blinded, randomized cross over trial will be consenting critical care trainees from the MCCTP at UPMC(Appendix 1 for consent forms). All participants will have similar baseline education in basic airway management, management of cardiovascular emergencies, and difficult airway management before testing occurs. Further, each participant will have similar clinical experience as a critical care trainee participating in METS at UPMC.

Each participant will undergo baseline testing using HST . Using 4 simulated clinical scenarios using the human simulator will test each participant. Participants will then be randomized into two groups. Control group (A) will receive no further training, while the intervention group ( B) will receive HST curriculum for medical crisis management. The groups will then be tested again after an interval of 1 month using 4 different simulated clinical scenarios. The groups will then be crossed over. The original control group (A) will now receive HST and the original intervention group ( B) will receive no further training. These two groups will again be tested using a third new set of simulated clinical scenarios. This study design is summarized in Appendix 2.

Both testing and the intervention will occur at the Peter Winter Institute for Simulation, Education and Research (WISER Center). All instructors and evaluators will be critical care faculty or senior fellows who have undergone training at WISER and are familiar with simulation teaching and evaluation.

The four medical crisis scenarios used for testing are designed to represent the most common medical crises experienced at UPMC. Each scenario will be programmed into the Laerdal SimMan human simulator. The basic physiologic problem and expected responses will be the same for all participants and all phases of testing; however, the scripted presentation will be varied to prevent pattern recognition. Participant performance will be evaluated using a checklist of expected actions as determined by the investigators. Each item will represent a communication skill, cognitive skill or a psychomotor skill. A total score as well as domain specific scores will be recorded at the end of each testing session for each participant. Blinded evaluators will perform all evaluations.

The intervention for this study will be a HST Curriculum. The curriculum will consist of two parts. One is a didactic review of crisis management principles. The second part is a simulation-based curriculum consisting of two scenarios. Each participant will undergo both scenarios and receive immediate feedback regarding their communication, cognitive and psychomotor performance.

ELIGIBILITY:
Inclusion Criteria:

* All consenting adult critical care medicine trainees at the MCCTP

Exclusion Criteria:

* Academic probation within training program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To assess the effectiveness of Human Simulation Training (HST) as an educational tool for teaching medical crisis management through objective measures of performance in the domains of communication, leadership, cognition and psychomotor skills. | 6 week intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh Venkataraman, MD, Principal Investigator — Department of Critical Care Mediine, University of Pittsburgh Medical Center; Lillian L Emlet, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Presbyterian Hospital, Pittsburgh, Pennsylvania, United States